CLINICAL TRIAL: NCT03722238
Title: MULTICENTER ACTUAL USE AND COMPLIANCE STUDY OF IBUPROFEN 600 MG IMMEDIATE RELEASE/EXTENDED RELEASE TABLETS AMONG TARGETED (AT-RISK) CONSUMERS IN A SIMULATED OVER-THE-COUNTER ENVIRONMENT
Brief Title: Actual Use and Compliance Study Of Ibuprofen 600 Mg Immediate Release/Extended Release Tablets In At-Risk OTC Consumers
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated on 18NOV2020 after an FDA meeting where it was determined no further actual use data was needed. There were no safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B4371011; MARATHON AUT (Other: Alias Study Number)
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Results first posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: The Actual Use Trial (AUT) design utilizes a real world setting to assess the ability of consumers to use an investigational product that will be marketed in an over-the-counter setting according to the proposed product labelling. The primary objective of this AUT is to evaluate compliance with the labeled dosing directions for Advil 12 Hour and to understand why misuse occurred and if it was a conscious decision by the subject. A secondary objective is to evaluate the safety of Advil 12 Hour in unsupervised actual use and how it relates to misuse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ibuprofen 600 mg Immediate Release/Extended Release Tablets (Experimental): Ibuprofen 600 mg Immediate Release/Extended Release Tablets
  Interventions: Drug: Ibuprofen 600 mg Immediate Release/Extended Release Caplet

INTERVENTIONS:
Drug: Ibuprofen 600 mg Immediate Release/Extended Release Caplet — Ibuprofen 600 mg Immediate Release/Extended Release Tablet to be adminstered orally (i.e., one caplet every 12 hours, not to exceed 2 caplets per day) for pain.

SUMMARY:
This will be an open-label, multicenter, 30-day, unsupervised AUS among targeted (at-risk) adult and adolescent consumers designed to mimic an OTC-like environment. More specifically, "at-risk" consumers, as discussed with the FDA, will comprise elderly consumers (>65 years of age), consumers with an increased risk of gastrointestinal (GI) bleeding or cardiovascular (CV) adverse events, consumers who experience severe pain, low literacy subjects, and adolescents (12-17 years of age). The total number of subjects expected to enroll into the study is approximately 820. Sites will be pharmacies in diverse geographic locations around the US. Prospective adult subjects will be recruited via general population and targeted risk condition advertising (although participants will not be informed as to specific health conditions for which they are being recruited), while adolescents will be recruited using targeted, outbound pre-recruiting telephone calls. Subjects (or the parents/guardians of prospective adolescent subjects) responding to the advertisements or recruitment calls will be initially screened by telephone, and eligibility will subsequently be verified in-person at the pharmacy site.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Male or female 18 years of age or older, has history of using oral OTC analgesics at OTC dose levels, defined as taking at least 5 doses/month on average during the past 3 months, and qualifies for inclusion in at least one risk group category, including cardiovascular, gastrointestinal bleeding, history of severe pain (≥5 episodes in last month) or >65 years of age (see Groups 1 4 in Section 3.1).

   OR Male or female 12-17 years of age and has history of using oral OTC analgesics at OTC dose levels, defined as taking at least 5 doses/month on average during the past 3 months.
2. Evidence of a personally signed and dated informed consent document (ICD), and in the case of minor adolescent subjects (12-17 years of age or adolescent subjects residing in states where the age of majority is > than 18), an assent document, indicating that the subject and where applicable a legally acceptable representative/parent(s)/legal guardian has been informed of all pertinent aspects of the study.
3. Willing and able to comply with scheduled visits, treatment plan, and other study procedures.
4. Willing (or in the case of adolescent subjects, the parent/guardian is willing) and able to purchase study medication.
5. Agrees the product purchased is for subject's own use and not to be shared.
6. Willing (or in the case of adolescent subjects, the parent/guardian is willing) and able to provide contact information for follow up purposes.

Exclusion Criteria

Subjects with any of the following characteristics/conditions will not be included in the study:

1. Subject (or parent/guardian, if applicable) cannot read, speak, and/or understand English.
2. Trained or employed as a healthcare professional.
3. Subject or someone else in the household is employed by a pharmaceutical company, medical practice or hospital, pharmacy, managed care or health insurance organization or a contract research organization.
4. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or potential subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
5. Participation in other studies involving investigational drug(s) within 6 months prior to study entry and/or during study participation.
6. Known hypersensitivity to ibuprofen, aspirin, or any other NSAIDs.
7. Subjects with the following clinical conditions which place them at excessively high risk or have ≥20% 10 year risk for atherosclerotic cardiovascular disease (ASCVD), as defined by the 2013 ACC/AHA Guidelines on the Assessment of Atherosclerotic Cardiovascular Risk, will not be included in the study: clinically established coronary heart disease; cerebrovascular disease; peripheral artery disease; abdominal aortic aneurysm; and chronic kidney disease. Subjects who have experienced a prior non fatal cardiovascular disease event (angina, heart failure, heart disease, heart attack, stroke/transient ischemic attack) or have had heart surgery or who currently have uncontrolled high blood pressure (either by self report or by measured systolic blood pressure higher than 180 mmHg or diastolic pressure higher than 120 mmHg at the time of the enrollment interview), will also be excluded from the study.
8. Subjects with concurrent or recent (within 30 days) use of anticoagulants, a prior history of complicated peptic ulcer, or a gastrointestinal bleeding event requiring hospitalization or blood transfusion.
9. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product (IP) administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
10. Pregnant female subjects; breastfeeding female subjects; and male and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for 28 days after the end of their 30-Day Use Phase or, for subjects who use the investigational product after Day 30, 28 days after the last recorded dose of investigational product.
11. 18 years of age or older and classified as normal literacy (REALM Test score ≥61) after the normal literacy group quotas (approximately 70% of adult subjects) are full or refuses to complete the REALM Test (note there is no corresponding literacy exclusion criterion for adolescent subjects based on REALM Teen score).
12. 18 years of age or older and classified as moderate (less frequent) oral OTC pain reliever user (<30 doses per month on average in the preceding 3 months) after the moderate user group quotas (approximately 33% of adult subjects) are full.
13. Not capable of swallowing a vitamin sized tablet.
14. Refuses to participate in required assessments (such as urine pregnancy, finger stick cholesterol or blood pressure tests, or unable or unwilling to comply with electronic diary procedures).

    The following additional exclusion criteria will be applied for adolescent subjects only (12-17 years of age):
15. Has developmental or learning disabilities that, in the judgment of the parent/guardian or the investigator, would interfere with study participation.
16. Another adolescent child from the family is already enrolled into the study, or parent/guardian does not agree that only one adolescent child from the family or household will be enrolled into the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- United States (27):
  - Mills Pharmacy at Bluff Park, Hoover, Alabama
  - Community Clinical Pharmacy, Mesa, Arizona
  - ACACIA Apothecary and Wellness, Tucson, Arizona
  - Coconut Grove Pharmacy, Miami, Florida
  - Summerfield Pharmacy, Riverview, Florida
  - Huff's Drug Store, Ellijay, Georgia
  - Family Care Pharmacy, Highland, Illinois
  - Rice's Pharmacy, Beaver Dam, Kentucky
  - Catonsville Pharmacy, Catonsville, Maryland
  - Goodrich Pharmacy, Anoka, Minnesota
  - Kemper Corner Drug, Elk River, Minnesota
  - Cub Pharmacy #744, Rosemount, Minnesota
  - The Medicine Shoppe and Elsberry Pharmacy, Elsberry, Missouri
  - Albers Medical Pharmacy, Kansas City, Missouri
  - Countryside Pharmacy, Savannah, Missouri
  - Texas Road Pharmacy, Monroe, New Jersey
  - Dakota Pharmacy of Bismarck, Bismarck, North Dakota
  - Family Prescription Center, Bethlehem, Pennsylvania
  - RxXPress Health Mart Pharmacy, Grove City, Pennsylvania
  - Medical Center Compounding Pharmacy & Health Center, Cleveland, Tennessee
  - Buckeye Drugs, Lebanon, Tennessee
  - Summerwood Pharmacy and Compounding, Houston, Texas
  - The Medicine Shoppe #708, Sherman, Texas
  - BrickStreet Pharmacy, Tyler, Texas
  - Bountiful Drug, Bountiful, Utah
  - The Medicine Center, Salt Lake City, Utah
  - Montpelier Pharmacy, Inc., Montpelier, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B4371011

RESULTS

PARTICIPANT FLOW:
Groups:
- Adult Compliance-Evaluable Population: The participants included in this group were male or female of age greater than or equal to (>=) 18 years at the time of enrollment with a history of using oral over-the-counter (OTC) analgesics at a dose levels of taking at least 5 doses per month on average during the past 3 months. Also, these participants had at least one of the following condition among cardiovascular risk, gastrointestinal bleeding risk, history of severe pain (>=5 episodes in last month) or >65 years of age. Participants were observed for the appropriate use of orally administered ibuprofen 600 milligram (mg) immediate release/extended release (IR/ER) tablets and compliance with the dosing instructions of total daily dose =1200 mg throughout the 30 days use.
- Adolescent Users: The participants were male or female with age between 12 to 17 years at the time of enrollment who had a history of using oral OTC analgesics at a dose levels of taking at least 5 doses per month on average during the past 3 months were observed for the appropriate use of orally administered ibuprofen 600 mg IR/ER tablets and compliance with the dosing instructions of total daily dose =1200 mg throughout the 30 days use.
Period: Overall Study
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Started | 608 | 5
Safety Set | 198 | 5
Actual Drug Users | 179 | 5
Completed (Completed=Participants for whom data collection was complete before early termination of the study.) | 143 | 4
Not Completed | 465 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 6 | 0
Not completed — Partial missing data | 44 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Other | 4 | 0
Not completed — Not returned to sign consent, download electronic diary application or to purchase study medication | 2 | 0
Not completed — Did not meet risk classification group criteria | 90 | 0
Not completed — Did not sign consent | 17 | 0
Not completed — Other eligibility criteria not met pre-consent | 22 | 0
Not completed — Not willing to purchase study medication | 142 | 0
Not completed — Did not qualify at re-screening and medical conditions | 133 | 0

BASELINE CHARACTERISTICS:
Population: Safety set included all the participants who signed informed consent and purchased the product.
Groups:
- Adult Compliance-Evaluable Population: The participants included in this group were male or female of age >=18 years at the time of enrollment with a history of using oral OTC analgesics at a dose levels of taking at least 5 doses per month on average during the past 3 months. Also, these participants had at least one of the following condition among cardiovascular risk, gastrointestinal bleeding risk, history of severe pain (>=5 episodes in last month) or >65 years of age. Participants were observed for the appropriate use of orally administered ibuprofen 600 mg IR/ER tablets and compliance with the dosing instructions of total daily dose =1200 mg throughout the 30 days use.
- Total: Total of all reporting groups
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users | Total
Number analyzed (Participants) | 198 | 5 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 5 | 5
  Between 18 and 65 years | 150 | 0 | 150
  >=65 years | 48 | 0 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 4 | 141
  Male | 61 | 1 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 1 | 11
  Not Hispanic or Latino | 188 | 4 | 192
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Data Analysis Set 1 Exceeding the Maximum Daily Dose of 1200 mg on 2 or More Calendar Days During the Use Period
Description: Use period was defined as 30 days from purchase.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: Participants who took at least 1 dose of study medication and recorded it in the electronic diary. Data analysis set 1 included the original data exactly as recorded by participants into their electronic diary.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 10.6 [6.1 to 15.1] | 0.0 [0.0 to 0.0]

2. Primary Outcome: Percentage of Participants in Data Analysis Set 2 Exceeding the Maximum Daily Dose of 1200 mg on 2 or More Calendar Days During the Use Period
Description: Use period was defined as 30 days from purchase.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: Participants who took at least 1 dose of study medication and recorded it in the electronic diary. Data analysis set 2 included the data clarified by the nurses during the end-of-study (EOS) interview under very specific pre-specified conditions when participants spontaneously identified dosing occasion specific entry errors in their original electronic diary data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 7.8 [3.9 to 11.8] | 0.0 [0.0 to 0.0]

3. Primary Outcome: Percentage of Participants in Data Analysis Set 3 Exceeding the Maximum Daily Dose of 1200 mg on 2 or More Calendar Days During the Use Period
Description: Use period was defined as 30 days from purchase.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: Participants who took at least 1 dose of study medication and recorded it in the electronic diary. Data analysis set 3 included the corrected/mitigated data that comprised of data analysis set 2 and misuses mitigated for additional diary entries judged to be incorrect or impossible based on participant's clear verbatim responses in the EOS interview.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 7.3 [3.5 to 11.1] | 0.0 [0.0 to 0.0]

4. Primary Outcome: Percentage of Participants in Data Analysis Set 4 Exceeding the Maximum Daily Dose of 1200 mg on 2 or More Calendar Days During the Use Period
Description: Use period was defined as 30 days from purchase.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: Participants who took at least 1 dose of drug and recorded in electronic diary. Data analysis set 4 included set 3 plus pre-specified mitigation factors (healthcare practitioner consultation, participants indicated: they would have taken opioid or other prescribed analgesic if not taken another dose, misuse of acetaminophen or other OTC analgesics and re-dosed earlier due to scheduling restrictions to prevent pain from returning) resulting in reclassification of misuses to acceptable status.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 2.8 [0.4 to 5.2] | 0.0 [0.0 to 0.0]

5. Secondary Outcome: Percentage of Participants in Data Analysis Set 1 Exceeding the Maximum Daily Dose of 1200 mg on 1 or More Calendar Days During the Use Period
Description: Use period was defined as 30 days from purchase.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 22.9 [16.7 to 29.1] | 0.0 [0.0 to 0.0]

6. Secondary Outcome: Percentage of Participants in Data Analysis Set 2 Exceeding the Maximum Daily Dose of 1200 mg on 1 or More Calendar Days During the Use Period
Description: Use period was defined as 30 days from purchase.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: Participants who took at least 1 dose of study medication and recorded it in the electronic diary. Data analysis set 2 included the data clarified by the nurses during the EOS interview under very specific pre-specified conditions when participants spontaneously identified dosing occasion specific entry errors in their original electronic diary data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 16.2 [10.8 to 21.6] | 0.0 [0.0 to 0.0]

7. Secondary Outcome: Percentage of Participants in Data Analysis Set 3 Exceeding the Maximum Daily Dose of 1200 mg on 1 or More Calendar Days During the Use Period
Description: Use period was defined as 30 days from purchase.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 14.0 [8.9 to 19.0] | 0.0 [0.0 to 0.0]

8. Secondary Outcome: Percentage of Participants in Data Analysis Set 4 Exceeding the Maximum Daily Dose of 1200 mg on 1 or More Calendar Days During the Use Period
Description: Use period was defined as 30 days from purchase.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 6.1 [2.6 to 9.7] | 0.0 [0.0 to 0.0]

9. Secondary Outcome: Percentage of Participants in Data Analysis Set 1 Exceeding the Maximum Daily Dose of 1200 mg on 1 or More Calendar Days During Use Period Due to Unintentional Misuse
Description: Unintentional misuse: Participants who did not understand the dosing instructions on the package. Use period was defined as 30 days from purchase.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 3.4 [0.7 to 6.0] | 0.0 [0.0 to 0.0]

10. Secondary Outcome: Percentage of Participants in Data Analysis Set 2 Exceeding the Maximum Daily Dose of 1200 mg on 1 or More Calendar Days During Use Period Due to Unintentional Misuse
Description: as for outcome 9
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 2.2 [0.1 to 4.4] | 0.0 [0.0 to 0.0]

11. Secondary Outcome: Percentage of Participants in Data Analysis Set 3 Exceeding the Maximum Daily Dose of 1200 mg on 1 or More Calendar Days During Use Period Due to Unintentional Misuse
Description: as for outcome 9
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 2.2 [0.1 to 4.4] | 0.0 [0.0 to 0.0]

12. Secondary Outcome: Percentage of Participants in Data Analysis Set 4 Exceeding the Maximum Daily Dose of 1200 mg on 1 or More Calendar Days During Use Period Due to Unintentional Misuse
Description: as for outcome 9
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 2.2 [0.1 to 4.4] | 0.0 [0.0 to 0.0]

13. Secondary Outcome: Percentage of Participants in Data Analysis Set 1 Exceeding the Maximum Amount Per Dose of 600 mg on 1 or More Occasions
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 30.7 [24.0 to 37.5] | 20.0 [0.0 to 55.1]

14. Secondary Outcome: Percentage of Participants in Data Analysis Set 2 Exceeding the Maximum Amount Per Dose of 600 mg on 1 or More Occasions
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 22.3 [16.2 to 28.4] | 20.0 [0.0 to 55.1]

15. Secondary Outcome: Percentage of Participants in Data Analysis Set 3 Exceeding the Maximum Amount Per Dose of 600 mg on 1 or More Occasions
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 19.0 [13.2 to 24.7] | 20.0 [0.0 to 55.1]

16. Secondary Outcome: Percentage of Participants in Data Analysis Set 4 Exceeding the Maximum Amount Per Dose of 600 mg on 1 or More Occasions
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 13.4 [8.4 to 18.4] | 0.0 [0.0 to 0.0]

17. Secondary Outcome: Percentage of Participants in Data Analysis Set 1 Exceeding the Maximum Amount Per Dose of 600 mg on 2 or More Occasions
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 17.9 [12.3 to 23.5] | 0.0 [0.0 to 0.0]

18. Secondary Outcome: Percentage of Participants in Data Analysis Set 2 Exceeding the Maximum Amount Per Dose of 600 mg on 2 or More Occasions
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 14.5 [9.4 to 19.7] | 0.0 [0.0 to 0.0]

19. Secondary Outcome: Percentage of Participants in Data Analysis Set 3 Exceeding the Maximum Amount Per Dose of 600 mg on 2 or More Occasions
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 13.4 [8.4 to 18.4] | 0.0 [0.0 to 0.0]

20. Secondary Outcome: Percentage of Participants in Data Analysis Set 4 Exceeding the Maximum Amount Per Dose of 600 mg on 2 or More Occasions
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 7.8 [3.9 to 11.8] | 0.0 [0.0 to 0.0]

21. Secondary Outcome: Percentage of Participants in Data Analysis Set 1 Exceeding the Maximum Daily Dose of 1200 mg on 10 or More Calendar Days
Description: Participants did not need to necessarily use the study medication for 10 consecutive days.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 1.1 [0.0 to 2.7] | 0.0 [0.0 to 0.0]

22. Secondary Outcome: Percentage of Participants in Data Analysis Set 2 Exceeding the Maximum Daily Dose of 1200 mg on 10 or More Calendar Days
Description: Participants did not need to necessarily use the study medication for 10 consecutive days.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 1.1 [0.0 to 2.7] | 0.0 [0.0 to 0.0]

23. Secondary Outcome: Percentage of Participants in Data Analysis Set 3 Exceeding the Maximum Daily Dose of 1200 mg on 10 or More Calendar Days
Description: Participants did not need to necessarily use the study medication for 10 consecutive days.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 1.1 [0.0 to 2.7] | 0.0 [0.0 to 0.0]

24. Secondary Outcome: Percentage of Participants in Data Analysis Set 4 Exceeding the Maximum Daily Dose of 1200 mg on 10 or More Calendar Days
Description: Participants did not need to necessarily use the study medication for 10 consecutive days.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

25. Secondary Outcome: Percentage of Participants in Data Analysis Set 1 Exceeding the Maximum Daily Dose of 1200 mg on 7 or More Calendar Days
Description: Participants did not need to necessarily use the study medication for 7 consecutive days.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 1.1 [0.0 to 2.7] | 0.0 [0.0 to 0.0]

26. Secondary Outcome: Percentage of Participants in Data Analysis Set 2 Exceeding the Maximum Daily Dose of 1200 mg on 7 or More Calendar Days
Description: Participants did not need to necessarily use the study medication for 7 consecutive days.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 1.1 [0.0 to 2.7] | 0.0 [0.0 to 0.0]

27. Secondary Outcome: Percentage of Participants in Data Analysis Set 3 Exceeding the Maximum Daily Dose of 1200 mg on 7 or More Calendar Days
Description: Participants did not need to necessarily use the study medication for 7 consecutive days.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 1.1 [0.0 to 2.7] | 0.0 [0.0 to 0.0]

28. Secondary Outcome: Percentage of Participants in Data Analysis Set 4 Exceeding the Maximum Daily Dose of 1200 mg on 7 or More Calendar Days
Description: Participants did not need to necessarily use the study medication for 7 consecutive days.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 0.6 [0.0 to 1.7] | 0.0 [0.0 to 0.0]

29. Secondary Outcome: Percentage of Participants in Data Analysis Set 1 Who Took More Than 2 Doses on a Calendar Day
Description: More than 2 doses on a calendar day means more than 2 dosing occasions on a calendar day.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 11.7 [7.0 to 16.4] | 0.0 [0.0 to 0.0]

30. Secondary Outcome: Percentage of Participants in Data Analysis Set 2 Who Took More Than 2 Doses on a Calendar Day
Description: More than 2 doses on a calendar day means more than 2 dosing occasions on a calendar day.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 7.8 [3.9 to 11.8] | 0.0 [0.0 to 0.0]

31. Secondary Outcome: Percentage of Participants in Data Analysis Set 3 Who Took More Than 2 Doses on a Calendar Day
Description: More than 2 doses on a calendar day means more than 2 dosing occasions on a calendar day.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 7.3 [3.5 to 11.1] | 0.0 [0.0 to 0.0]

32. Secondary Outcome: Percentage of Participants in Data Analysis Set 4 Who Took More Than 2 Doses on a Calendar Day
Description: More than 2 doses on a calendar day means more than 2 dosing occasions on a calendar day.
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 2.8 [0.4 to 5.2] | 0.0 [0.0 to 0.0]

33. Secondary Outcome: Percentage of Participants in Data Analysis Set 1 Who Re-dosed in Less Than (<)12 Hours, <10 Hours and <8 Hours on 1 or More Occasions
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants
  Re-dosed in <12 Hours | 47.5 [40.2 to 54.8] | 0.0 [0.0 to 0.0]
  Re-dosed in <10 Hours | 36.3 [29.3 to 43.4] | 0.0 [0.0 to 0.0]
  Re-dosed in <8 Hours | 29.1 [22.4 to 35.7] | 0.0 [0.0 to 0.0]

34. Secondary Outcome: Percentage of Participants in Data Analysis Set 2 Who Re-dosed in Less Than (<)12 Hours, <10 Hours and <8 Hours on 1 or More Occasions
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants
  Re-dosed in <12 Hours | 43.0 [35.8 to 50.3] | 0.0 [0.0 to 0.0]
  Re-dosed in <10 Hours | 28.5 [21.9 to 35.1] | 0.0 [0.0 to 0.0]
  Re-dosed in <8 Hours | 19.6 [13.7 to 25.4] | 0.0 [0.0 to 0.0]

35. Secondary Outcome: Percentage of Participants in Data Analysis Set 3 Who Re-dosed in Less Than (<)12 Hours, <10 Hours and <8 Hours on 1 or More Occasions
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants
  Re-dosed in <12 Hours | 42.5 [35.2 to 49.7] | 0.0 [0.0 to 0.0]
  Re-dosed in <10 Hours | 26.8 [20.3 to 33.3] | 0.0 [0.0 to 0.0]
  Re-dosed in <8 Hours | 17.3 [11.8 to 22.9] | 0.0 [0.0 to 0.0]

36. Secondary Outcome: Percentage of Participants in Data Analysis Set 4 Who Re-dosed in Less Than (<)12 Hours, <10 Hours and <8 Hours on 1 or More Occasions
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants
  Re-dosed in <12 Hours | 39.7 [32.5 to 46.8] | 0.0 [0.0 to 0.0]
  Re-dosed in <10 Hours | 18.4 [12.8 to 24.1] | 0.0 [0.0 to 0.0]
  Re-dosed in <8 Hours | 12.3 [7.5 to 17.1] | 0.0 [0.0 to 0.0]

37. Secondary Outcome: Percentage of Participants in Data Analysis Set 1 Who Used the Product on More Than 10 Consecutive Calendar Days
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 22.3 [16.2 to 28.4] | 0.0 [0.0 to 0.0]

38. Secondary Outcome: Percentage of Participants in Data Analysis Set 2 Who Used the Product on More Than 10 Consecutive Calendar Days
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 22.9 [16.7 to 29.1] | 0.0 [0.0 to 0.0]

39. Secondary Outcome: Percentage of Participants in Data Analysis Set 3 Who Used the Product on More Than 10 Consecutive Calendar Days
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 179 | 5
Percentage of participants | 22.9 [16.7 to 29.1] | 0.0 [0.0 to 0.0]

40. Secondary Outcome: Percentage of Participants in Data Analysis Set 4 Who Used the Product on More Than 10 Consecutive Calendar Days
Time Frame: From first purchase of study drug (Day 1) to Day 30
Population: Data for this outcome measure was not estimable based on the pre-specified mitigation factors, as consecutive use days were not dosing errors and therefore not mitigable. Hence, no results were calculated.
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: First purchase of study drug up to maximum of 45 days after last dose of study drug (for up to 75 days)
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety set included all the participants who signed informed consent and purchased the product.
Arm/Group | Adult Compliance-Evaluable Population | Adolescent Users
All-Cause Mortality (participants affected / at risk) | 1/198 | 0/5
Serious Adverse Events (participants affected / at risk) | 4/198 | 0/5
Other Adverse Events (participants affected / at risk) | 9/198 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adult Compliance-Evaluable Population (N=198) | Adolescent Users (N=5)
Victim of crime (Social circumstances) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Death (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adult Compliance-Evaluable Population (N=198) | Adolescent Users (N=5)
Nasopharyngitis (Infections and infestations) | 5 | 0
Nausea (Gastrointestinal disorders) | 4 | 1

LIMITATIONS AND CAVEATS:
This study was terminated early due to recruitment problems and challenges. No safety concerns led to the decision to terminate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT03722238/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT03722238/SAP_001.pdf